CLINICAL TRIAL: NCT01275560
Title: Does the Negativation of the Glucose Hydrogen Breath Test Come Along With a Reduction of the Symptoms of Gaz Incontinence ?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008/073/HP
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Anal Incontinence
MeSH Terms: conditions — Encopresis | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metronidazole (Experimental): 3 intakes per day during 10 days
  Interventions: Drug: Metronidazole
- Carbosylane (Active Comparator): 3 intakes per daysduring 10 days
  Interventions: Drug: CArbosylane

INTERVENTIONS:
Drug: Metronidazole — Metronidazole,per os,500mg, 3 per day during 10 days
  Arms: Metronidazole
Drug: CArbosylane
  Arms: Carbosylane

SUMMARY:
The objectives of this work are: 1/to estimate the frequency of a positive glucose breath test in favour of a small intestinal bacterial overgrowth in a population of patients consulting for gaz incontinence by comparison to a population of control subjects; 2/to estimate versus a conventional treatment the efficiency of an antibiotic treatment; in case of small intestinal bacterial overgrowth diagnosed by the glucose breath test, to improve gaz incontinence

ELIGIBILITY:
Inclusion Criteria:

* Gaz incontinence for more than 3 months
* Afflilied to national health security
* Having read and sign the information letter and consent form

Exclusion Criteria:

* Pregnancy
* use of antibiotics, probiotics, IPP for less tha n 3 months
* past of small intestinal bacterial overgrowth
* ischemic, inflammatory colitis,colo-rectal cancer
* diabetes
* allergy to metronidazole
* psychiatric disease
* patients who do not speak or read french

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
number of gaz incontinence episodes | 3 days before randomization and treatement and 3 days after 10 days of treatment (antibiotic or conventionnal treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Physiology Unit, Hopital Charles Nicolle, 1 rue de Germont, Rouen, France